CLINICAL TRIAL: NCT05475496
Title: Quality of Life of Elderly Cardiac Patients With Multimorbidity and Prevalence of Burnout Among Their Caregivers in Sohag Governorate
Brief Title: Quality of Life of Elderly Patients and Burnout Among Their Care Givers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shimaa Harris Ahmed, Assistant lecturer of public health and community medicine, faculty of medicine, sohag university, Sohag University
Other Study IDs: Soh-Med-22-06-15
Record Dates: First submitted 2022-07-22; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Elderly Cardiac Patients With Multimorbidity and Burnout Among Their Caregivers

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Elderly cardiac patients with multimorbidity and their caregivers: elderly patients (60 years and over) [2] with multimorbid conditions and a cardiovascular disease is one of them .
  caregivers of elderly patients included in the study
  Interventions: Other: Measurements of quality of life and burnout

INTERVENTIONS:
Other: Measurements of quality of life and burnout — WHOQOL-Bref questionnaire to assess the health related quality of life of the elderly cardiac patients. WHOQOL-Bref assesses Physical health (7 items), Psychological health (6 items), Social relationships (3 items) and the environment ( 8 items ), in addition to two items asking about overall perception of life and general health. Items are rated on a 5 point ordinal scale, domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life).
  Maslach Burnout Inventory questionnaire to measure burnout among caregivers, it includes 3 components: emotional exhaustion (9 items), depersonalization(5items) and personal accomplishment(8 items).

SUMMARY:
Older people with multimorbidity are frequent users of health care services, and there is a relationship between the number of chronic conditions and health care costs. In addition, multimorbidity increases the risk of mortality and functional decline, and this negatively impacts health-related quality of life

. Furthermore, research tends to focus on individual organ systems, often ignoring the complexity of care for older people with multimorbidity. Moreover, patient QoL is a meaningful measure in the evaluation of health care services and patient-reported outcome Caregiving demands significantly reduce caregivers' opportunities to have a lifestyle in which leisure or time for themselves is available. According to different empirically supported theoretical frameworks that point to the importance for caregivers of experiencing pleasant events and receiving positive reinforcement in their daily lives in order to maintain a positive mood, not engaging in personally satisfying activities may result in more social withdrawal and depression, putting caregivers at risk of developing emotional disorders.

DETAILED DESCRIPTION:
As the percentage of elderly cardiac population is growing and most of them have multimorbid conditions, we should find ways to improve their of life and to avoid their caregivers being burned out.

Asses quality of life of cardiac elderly patients with multimorbidity and to investigate the prevalence of burnout among their caregivers This study of multimorbidity among elderly cardiac patients attending Sohag university cardiac outpatient clinic and burnout among their care givers aims to:-

1. Study the effect of multimorbidity on health related quality of life of elderly cardiac patients.
2. Study determinants of health related quality of life among elderly cardiac patients with multimorbidity.
3. Study burnout prevalence among care givers

ELIGIBILITY:
Inclusion Criteria:

* elderly patients (60 years and over) [2] with multimorbid conditions and a cardiovascular disease is one of them .

caregivers of elderly patients included in the study.

Exclusion Criteria:

* patients and caregivers who will refuse to participate in this study and patients with disturbed conscious level and mentally disabled.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Elderly patients with multimorbidity attending cardiac out patient clinic in Sohag University hospital and their caregivers
Sampling Method: Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life of elderly patients | 6 months
  Measuring the quality of life of elderly patients with cardiovascular and other morbid conditions using WHOQOL-Bref questionnaire
Burnout among caregivers | 6 months
  Measuring the prevalence of burnout among caregivers using Maslach Burnout Inventory questionnaire